CLINICAL TRIAL: NCT03512717
Title: A Multi-center, Randomized, Subject-evaluator Blind, Active Controlled Design Clinical Study to Determine the Efficacy and Safety of Potenfill for Temporary Penile Enhancement
Brief Title: Efficacy and Safety of Potenfill for Temporary Penile Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT05-KR17PGE308
Record Dates: First submitted 2018-04-27; First posted 2018-05-01 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Penile Enhancement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potenfill (Experimental)
  Interventions: Device: Potenfill
- Powerfill (Active Comparator)
  Interventions: Device: Powerfill

INTERVENTIONS:
Device: Potenfill — Maximum: 22ml
  Arms: Potenfill
Device: Powerfill — Maximum: 22ml
  Arms: Powerfill

SUMMARY:
The purpose of this study is to evlauate the efficacy and safety of poteinfill, compared to the powerfill.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged above 19 and below 65. (20≤male≥65)
2. be rating himself, when screening, as "Small or Very Small" on Self-Questioned Questionnaire ( SQQ) including the question: " How do you rate your penile size? // Very small, Small, Normal, Big, Very Big?"
3. Subjects will sign an informed consent form

Exclusion Criteria:

1. Prior treatment for penile enhancement (e.g. fat, dermal graft).
2. Subjects who have penile malformation (e.g. Peyronie's disease), which can make impossible to perform the intervention
3. Allergic to hyalluronic acid.
4. Inflammatory or/and infectious disease on penis that can affect on this study

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
the Penile Circumference difference at 24 weeks from baseline | 24 weeks
  Penile Circumference: The average of Distal-, Mid-, and Proximal-penis measurements when relaxed by tape measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Gangdong Sacred Heart Hospital, Hallym Univ, Seoul, South Korea